CLINICAL TRIAL: NCT06633497
Title: Evaluating the Role of the Microbiome in Antidepressant Treatment in Adolescents.
Status: Not yet recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: Rady Children's Hospital, San Diego (Other)
Responsible Party: Principal Investigator, Rob Knight, Professor, University of California, San Diego
Other Study IDs: 807323
Record Dates: First submitted 2024-10-03; First posted 2024-10-09 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Depression in Adolescence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn about the role of the human gut microbiome in antidepressant treatment response in adolescents with Major Depressive Disorder (MDD). Specifically, the study aims to collect microbiota samples of adolescents treated with fluoxetine, over the span of 8-weeks, to:

* determine the influence of the microbiome on the efficacy of fluoxetine to treat adolescent depression.
* test whether the gut microbiome from different timepoints can predict ultimate success of fluoxetine
* investigate the interaction of gut microbiome composition and pharmacogenetic metabolizer status on steady-state plasma concentrations of fluoxetine.

Depression symptom severity will be evaluated upon enrollment and 6-weeks into antidepressant treatment.

DETAILED DESCRIPTION:
For this project the investigators are interested in changes in the gut microbiome associated with adolescent depression and the influence of the microbiome on the efficacy of fluoxetine to treat adolescent depression. It is hypothesized that the composition of the human gut microbiome alters the response to fluoxetine of adolescents with depression. This study aims to collect gut microbiota of adolescents being treated with antidepressants at several timepoints to (1) determine the efficacy of fluoxetine to treat depression, (2) test whether the gut microbiome from different timepoints can predict ultimate success of fluoxetine, and (3) investigate the interaction of gut microbiome composition and pharmacogenetic metabolizer status on steady-state plasma concentrations of fluoxetine. Adolescent patients with clinically significant depressive symptoms who are prescribed fluoxetine, from Rady Children's Hospital San Diego (RCHSD) Inpatient Child and Adolescent Psychiatry Services (CAPS), will be recruited for this study. Up to twelve stool samples are planned to be collected, including prior to start of antidepressant treatment for a baseline measure of gut microbiome composition, daily samples over during the first week of fluoxetine treatment, and then biweekly collections until the end of the 8-week study duration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from all ethnic backgrounds will be eligible to participate.
* Having clinically significant depressive symptoms based on a score >40 on the Children's Depression Rating Scale-Revised
* Prescribed more than 5mg of Fluoxetine (Prozac)
* Has an identifiable legal guardian.

Exclusion Criteria:

* Has been taking a standing psychotropic medication in the past 6 months
* Has been taking antibiotics or metformin during the past 6 months (known strong effects on gut microbiome)
* Admitted to RCHSD CAPS post-overdose (potential strong effects on gut microbiome)
* Currently using nicotine-containing substances (known strong effects on gut microbiome)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescents ages 13-17 with depression diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome composition | Stool samples will be collected at enrollment (baseline), then following enrollment: daily for the first 7 days and biweekly at weeks 2, 4, 6, and 8.
  Gut microbiome composition will be characterized by analysis of stool samples
Efficacy of fluoxetine to treat depression symptoms in adolescents | The CDRS-R will be administered at baseline and week 6.
  Fluoxetine success will be characterized by change, from baseline to week 6 follow-up, of Children's Depression Rating Scale, Revised (CDRS-R) scores.

SECONDARY OUTCOMES:
Efficacy of fluoxetine to improve self-reported depression symptoms in adolescents | The MFQ will be administered at baseline and week 6.
  Fluoxetine success will be characterized by the change, from baseline to week 6 follow-up, of self-reported depression symptom severity indicated by Mood and Feelings Questionnaire (MFQ) scores.
Efficacy of fluoxetine to treat anxiety symptoms in adolescents | The SCARED will be administered at baseline and week 6.
  Fluoxetine success will be characterized by the change, from baseline to week 6 follow-up, of self-reported severity of recent anxiety symptoms indicated by the Screen for Child Anxiety Related Disorders (SCARED) scores.
Pharmacogenetic (PGx) metabolizer status | A saliva sample is collected for pharmacogenetic analysis at baseline
  Patients are divided into metabolic phenotype groups denoted as poor, intermediate, and ultrarapid metabolizers based on their specific variant profile of pharmacokinetic genes.
Steady-state plasma concentrations of fluoxetine | Sample collected at week 6
  Steady-state plasma sample concentrations of fluoxetine and (active metabolite norfluoxetine).

CONTACTS AND LOCATIONS:
Overall Officials: Rob Knight, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- Rady Children's Hospital San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No